CLINICAL TRIAL: NCT05329480
Title: Cardiac and Vascular Responses to Creatine Supplementation in Elderly Men
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radford University (Other)
Responsible Party: Principal Investigator, Adrian Aron, Professor, Radford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-431
Record Dates: First submitted 2022-03-07; First posted 2022-04-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Function and Hemodynamics
MeSH Terms: interventions — Creatine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Creatine Monohydrate Supplementation (Experimental): Blinded subjects are instructed to ingest 20g of creatine monohydrate for 7 days divided into 4 dosages of 5g each that should be taken with water or other liquids throughout the day (breakfast, lunch, afternoon and evening).
  Interventions: Dietary Supplement: Creatine Monohydrate
- Maltodextrin Supplementation (Placebo Comparator): Blinded subjects are instructed to ingest 20g of maltodextrin for 7 days divided into 4 dosages of 5g each that should be taken with water or other liquids throughout the day (breakfast, lunch, afternoon and evening).
  Interventions: Dietary Supplement: Maltodextrin
- Control (No Intervention): Participants in the control group do not receive a supplement (creatine or placebo) to ingest over the 7 day period.

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — Creatine Monohydrate powder, 4 separate 5g doses per day for 7 days.
  Arms: Creatine Monohydrate Supplementation
Dietary Supplement: Maltodextrin — Maltodextrin powder, 4 separate 5g doses per day for 7 days.
  Arms: Maltodextrin Supplementation

SUMMARY:
The purpose of this study is to investigate the impact of creatine supplementation alone or in combination with a moderate session of physical activity on vascular reactivity and heart hemodynamics in elderly men.

DETAILED DESCRIPTION:
Before beginning baseline testing, subjects' vitals will be measured (heart rate, blood pressure) in order to ensure that they are safe to participate in the submaximal exercise test. Subjects will also complete the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) to screen for cardiovascular risk factors. Information about physical activity level, medical history, and creatine supplementation use history will also be acquired. After anthropometric measurements, subjects will be asked to lay down in a hospital-type bed for measuring heart function and vascular responses at rest.

For measures of heart function, a non-invasive bioimpedance device will be used. Five ECG electrodes will be placed on chest and neck areas that will continuously collect information about heart rate, stroke volume, contractility index, ejection fraction and systemic vascular resistance. Vascular responses will be assessed using a non-invasive arterial pulse wave velocity equipment. This test uses four blood pressure cuffs placed on the wrists and calves, which, after 10 seconds inflation, are able to calculate an index of stiffness.

After resting values are collected, the cuffs will be removed, and subjects will be asked to walk on a treadmill at 6 km/h (3.1mph) and 5% grade for 10 minutes. During the treadmill walking, subjects will have their heart monitored using the non-invasive bioimpedance device with the ECG attached to their chest and neck. After 10 minutes have passed, subjects will be asked to step down from the treadmill and lay down on in the same hospital type bed.

At this time, the four blood pressure cuffs will be placed again on the wrists and calves to measure the vascular responses. We plan on performing two arterial stiffness measurements, after 10 and 20 minutes of the treadmill walking. After 20 minutes of monitoring while lying in bed, subjects will be disconnected from all ECGs and blood pressure cuffs.

Randomization in one of the three groups will occur using a computer generated sequence. The groups will have 15 subjects each and will consist of creatine supplementation, placebo supplementation (maltodextrin) and control (no supplementation). After randomization, subjects will receive their assigned packages containing the supplementation supplies corresponding to their group allocation (creatine or placebo). After 7 days of 20g/day supplementation, subjects will be asked to come back to the testing center for a repeat of the exercise test and corresponding heart monitoring and vascular responses before and after the treadmill walk.

To ensure good compliance with supplementation, subjects will receive daily text messages with reminders about their dose ingestion. The 20g/day will be divided in 4 dosages of 5g each that should be taken with water or other liquids throughout the day (breakfast, lunch, afternoon and evening).

ELIGIBILITY:
Inclusion Criteria:

* Males
* 55-80 years old
* No restrictions based on race, ethnicity, or socioeconomic status

Exclusion Criteria:

* Females
* <55 or >80 years old
* Individuals with known serious cardiac pathology
* Individuals with known serious kidney pathology
* Appropriate for moderate intensity exercise (screening using PAR-Q+)
* Individuals currently consuming or had consumed creatine supplement within 3 months prior to screening

Ages: 55 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in brachial-ankle pulse wave velocity (baPWV) | Baseline and day 8.
  PWV is a validated, non-invasive, clinical technique used to measure arterial stiffness. Participants will lay supine, and 4 blood pressure cuffs will be wrapped around the limbs. One cuff on each arm (brachial artery) and one cuff on each ankle (posterior tibial artery). The distance between the two sampling points (arms and ankles) will be calculated according to the height of the subject. PWV is measured as the distance between two recording sites divided by the transit time of the pulse wave detected. PWV will be given as meters/second. Values will be measured at rest, during a 10 minute bout of exercise, 10 and 20 minutes post-exercise.

SECONDARY OUTCOMES:
Stroke Volume | Baseline and day 8.
  Determined by bioimpedance. The technique measures the change in impedance using a high frequency alternating electrical current (66 kHz) of low magnitude (4.5 mA peak to peak) between different electrodes positioned around the chest and neck. Values will be measured at rest, during a 10 minute bout of exercise, 10 and 20 minutes post-exercise.
Cardiac Index | Baseline and day 8.
  Determined by bioimpedance. The technique measures the change in impedance using a high frequency alternating electrical current (66 kHz) of low magnitude (4.5 mA peak to peak) between different electrodes positioned around the chest and neck. Values will be measured at rest, during a 10 minute bout of exercise, 10 and 20 minutes post-exercise.
Systemic Vascular Resistance | Baseline and day 8.
  Determined by bioimpedance. The technique measures the change in impedance using a high frequency alternating electrical current (66 kHz) of low magnitude (4.5 mA peak to peak) between different electrodes positioned around the chest and neck. Values will be measured at rest, during a 10 minute bout of exercise, 10 and 20 minutes post-exercise.
Ejection Fraction | Baseline and day 8.
  Determined by bioimpedance. The technique measures the change in impedance using a high frequency alternating electrical current (66 kHz) of low magnitude (4.5 mA peak to peak) between different electrodes positioned around the chest and neck. Values will be measured at rest, during a 10 minute bout of exercise, 10 and 20 minutes post-exercise.
Contractility Index | Baseline and day 8.
  Determined by bioimpedance. The technique measures the change in impedance using a high frequency alternating electrical current (66 kHz) of low magnitude (4.5 mA peak to peak) between different electrodes positioned around the chest and neck. Values will be measured at rest, during a 10 minute bout of exercise, 10 and 20 minutes post-exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Carilion Roanoke Community Hospital, Roanoke, Virginia, United States

REFERENCES:
- [Derived] Aron A, Landrum EJ, Schneider AD, Via M, Evans L, Rawson ES. Effects of acute creatine supplementation on cardiac and vascular responses in older men; a randomized controlled trial. Clin Nutr ESPEN. 2024 Oct;63:557-563. doi: 10.1016/j.clnesp.2024.07.008. Epub 2024 Jul 22. PMID 39047868